CLINICAL TRIAL: NCT05543850
Title: Portable Artificial Pancreas Applied for Youth and Adolescents
Acronym: PAPAYA 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inreda Diabetic B.V. (Industry)
Collaborators: Stichting Robopump (Unknown); Rijnstate ziekenhuis (Unknown); Kinder Diabetes Centrum Nijmegen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL79829.000.22
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Intervention Model Description: The study is a monocenter, randomized cross-over trial. The total duration of the study will be three months: two weeks open loop control and 4-6 training days followed by a two-week closed-loop period, or vice versa, with at least 2 weeks in between.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open loop control (Active Comparator): In this arm, the patients will use their usual diabetes therapy. Additionally, patients will wear a blinded DexcomG6 for data collection during the open loop period.
  Interventions: Device: Open-loop control
- Bi-hormonal closed-loop control (Experimental): In this arm, treatment consists of the bi-hormonal closed-loop system. A short acting insulin analogue (Humalog, 3 ml pre-filled cartridge, Eli Lilly) and glucagon (Glucagen, Novo Nordisk; 3.15 ml cartridge Accu-Chek Spirit, Roche) will be administered according to the closed-loop algorithm. Additionally, patients will wear a blinded DexcomG6 for data collection during the closed loop period.
  Interventions: Device: Bi-hormonal closed-loop control

INTERVENTIONS:
Device: Bi-hormonal closed-loop control — During bi-hormonal closed-loop control insulin and glucagon are administered to the developed closed-loop algorithm. Aditionally, patients will wear a blinded Dexcom G6 for data collection during the closed loop period.
  Other Names: Artificial Pancreas (AP); bi-hormonal AP system; AP5
  Arms: Bi-hormonal closed-loop control
Device: Open-loop control — During open-loop control the patients will use their usual diabetes therapy. Aditionally, patients will wear a blinded Dexcom G6 for data collection during the open loop period.
  Arms: Open loop control

SUMMARY:
The purpose of this study is to determine the performance of a bi-hormonal reactive closed-loop system in adolscents with type 1 diabetes mellitus. The percentage of time spent in the target range (3.9-10.0 mmol/L) is the main outcome and will be compared between the bi-hormonal closed-loop system and the current treatment of the patients. Also, safety parameters, pharmacodynamics and patient reported outcomes (expectations, trust and treatment satisfaction scores) are compared.

This study is a monocenter, randomized, cross-over trial with 20 subjects. The subjects will be randomized to receive either the open-loop therapy or the closed-loop therapy for the first two-week study period and switch to the alternate treatment with at least two weeks in between.

DETAILED DESCRIPTION:
Background of the study:

Inreda Diabetic B.V. (Goor, The Netherlands) developed a bi-hormonal reactive closed loop system to automate glucose regulation (artificial pancreas; AP) in patients with diabetes mellitus type 1. In previous studies, we tested the performance and safety of this bi-hormonal closed-loop system in an outpatient setting in patients with type 1 diabetes mellitus (T1DM) for a duration up to 2 weeks, leading to CE-marking of the system. The device is currently intended for insulin-dependent adult patients with diabetes. However, there is great need to improve glycaemic control in youth and adolescents with diabetes.

Objective of the study:

The main objective of this study is to determine the performance of the closed-loop system in adolescents with T1DM. Secondary objectives include: to assess the safety of the closed-loop system; to determine the time that the closed-loop algorithm is active; and to assess expectations and treatment satisfaction of the closed-loop system.

Study design:

This study is a monocenter randomized cross-over trial.

Study population:

The study population will comprise 20 patients with T1DM, between 12 and 18 years old, not having impaired awareness of hypoglycaemia, and who are treated with insulin therapy for at least 6 months. Patients receiving treatment with multiple daily injections (MDI) or continuous subcutaneous insulin injections (CSII), and in addition glucose monitoring using self-monitored blood glucose (SMBG), flash glucose monitoring (FGM) or continuous glucose monitoring (CGM) are included into the study.

Intervention:

The intervention includes 2 weeks of closed-loop control with the artificial pancreas (AP) of Inreda Diabetic. The device uses 2 subcutaneous glucose sensors, 2 subcutaneous infusion sets, and incorporates 2 pumps and a reactive closed-loop algorithm. During 4-6 days before the intervention the patients receive training on the use of the closed-loop system and will start using the device under close supervision. The control arm (open loop treatment) consists of the patient's standard therapy at home for 2 weeks.

Main study parameters/endpoints:

Main study parameter is the percentage of time spent in the target range (3.9-10.0 mmol/L), which will be compared between the open and closed-loop periods for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes mellitus
* Twelve to eighteen years old;
* Treated with insulin therapy for at least 6 months;
* Willing and able to sign informed consent or to assent to study participation.

Exclusion Criteria:

* Impaired awareness of hypoglycaemia (score ≥ 4) according to Gold and/or Clarke questionnaire[6,7];
* BMI ≥ 35 kg/m2;
* Pregnancy and/or breastfeeding;
* HbA1c > 97 mmol/mol (11.0%);
* Use of acetaminophen (paracetamol) during the open loop or closed-loop period,as this may influence the sensor glucose measurements;
* Limited ability to see, hear or feel the alarm signals of the closed-loop system;
* Unwillingness to act in response to the alarm signals;
* Living alone during the night during the closed-loop period (the patient may ask someone to stay over temporarily);
* Expected poor internet connectivity regarding 24/7 tele monitoring;
* Any condition that the local investigator feels would interfere with trial participation or evaluation of the results.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Time in range | 2 weeks
  The proportion of time spent in the range of 3.9-10.0 mmol/L in %

SECONDARY OUTCOMES:
Time in hypoglycemia 1 | 2 weeks
  The proportion of time spent in hypoglycemia (<3.9 mmol/L) in %
Time in hypoglycemia 2 | 2 weeks
  The proportion of time spent in hypoglycemia (<3.0 mmol/L) in %
Time in hyperglycemia 1 | 2 weeks
  The proportion of time spent in hyperglycemia (>10.0 mmol/L) in %
Time in hyperglycemia 2 | 2 weeks
  The proportion of time spent in hyperglycemia (>13.9 mmol/L) in %
Mean glucose concentration | 2 weeks
  Mean glucose concentration in mmol/L
Median glucose concentration | 2 weeks
  Median glucose concentration in mmol/L
Glycemic variability - Coefficient of variation | 2 weeks
  Coefficient of variation (standard deviation divided by the mean) in %
Glycemic variability - Interquartile range | 2 weeks
  Interquartile range in mmol/L
Mean glucose concentration during the day | 2 weeks
  Mean glucose concentration in mmol/L during the day (6AM - 12PM)
Mean glucose concentration during the night (12PM - 6AM) | 2 weeks
  Mean glucose concentration in mmol/L during the night (12PM - 6AM)
Median glucose concentration during the day (6AM - 12PM) | 2 weeks
  Median glucose concentration in mmol/L during the day (6AM - 12PM)
Median glucose concentration during the night (12PM - 6AM) | 2 weeks
  Median glucose concentration in mmol/L during the night (12PM - 6AM)
Time spent in hypoglycemia during the night | 2 weeks
  Time spent in hypoglycemia (<3.9 mmol/L) during the night (12PM - 6AM) in %
Time spent in hyperglycemia during the night | 2 weeks
  Time spent in hyperglycemia (>10.0 mmol/L) during the night (12PM - 6AM) in %
Time spent in euglycemia during the night | 2 weeks
  Time spent in euglycemia (<3.9 mmol/L and <10 mmol/L) during the night (12PM - 6AM) in %
Time spent in hypoglycemia during the day | 2 weeks
  Time spent in hypoglycemia (<3.9 mmol/L) during the day (6AM - 12PM) in %
Time spent in hyperglycemia during the day | 2 weeks
  Time spent in hyperglycemia (>10.0 mmol/L) during the day (6AM - 12PM) in %
Time spent in euglycemia during the day | 2 weeks
  Time spent in euglycemia (<3.9 mmol/L and <10 mmol/L) during the day (6AM - 12PM) in %
Algorithm active time | 2 weeks
  Time that the closed-loop algorithm is active in %
Expectations | 2 weeks
  INSPIRE questionnaire (only for closed loop)
Trust | 2 weeks
  TAS questionnaire (only for closed loop)
Satisfaction | 2 weeks
  DTSQ questionnaire (for open loop and closed loop)

OTHER OUTCOMES:
Gender | Baseline
  Gender (M/F)
Weight | Baseline
  Weight in kg
Length | Baseline
  Length in cm
HbA1c plasma concentration | Baseline
  HbA1c plasma concentration in mmol/mol
Current medication use | Baseline
  List of medication names and corresponding dosages
Insulin dose | 2 weeks
  Daily average of insulin in units
Glucagon dose | 2 weeks
  Daily average of glucagon in units

CONTACTS AND LOCATIONS:
Overall Officials: Arianne Bon, MD, PhD, Principal Investigator — Rijnstate ziekenhuis
Locations (1):
- Rijnstate Ziekenhuis, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No